CLINICAL TRIAL: NCT05693259
Title: Improvement Effect of Functional Dyspepsia After Drinking Alkaline Ionized Water From Alkaline Ionizer in Functional Ddyspepsia Patients
Brief Title: Improvement of Functional Dyspepsia After Drinking Alkaline Ionized Water From Alkaline Ionizer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wonju Severance Christian Hospital (Other)
Responsible Party: Principal Investigator, Kyu Jae Lee, Professor, Wonju Severance Christian Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EMB-2022-01
Record Dates: First submitted 2022-12-08; First posted 2023-01-20 (Actual); Last update posted 2023-01-20 (Actual); Status verified 2023-01

CONDITIONS: Functional Dyspepsia

STUDY DESIGN:
Intervention Model Description: * Control group (PW): purified water-drinking group
  * Experimental group (EARW): Electrolyzed alkaline reduced water drinking group
Who Masked: Participant, Investigator
Masking Description: Double blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EARW group (Experimental): Patients in EARW group drink EARW (pH 9.5) 10 mL/kg body weight per a day using experimental device installed in the house for 6 weeks. We recommend to drink water in empty stomach three or four times a day. The water generated from device will be administered immediately, not to be stored.
  Interventions: Device: Electrolyzed Alkaline Reduced Water (EARW) generated from electrolyzed ionizer
- PW group (Sham Comparator): Patients in PW group drink PW (pH 9.5) 10 mL/kg body weight per a day using Sham device installed in the house for 6 weeks. We recommend to drink water in empty stomach three or four times a day. The water generated from device will be administered immediately, not to be stored. Sham device was built in the same shape and operation as the experimental device.
  Interventions: Device: Electrolyzed Alkaline Reduced Water (EARW) generated from electrolyzed ionizer

INTERVENTIONS:
Device: Electrolyzed Alkaline Reduced Water (EARW) generated from electrolyzed ionizer — Patient will be allocated randomly to two groups: EARW and PW groups. For 6 weeks, patients drink water (10mL/kg body weight/day ) generated from the device installed in the house before starting intervention. Patients will be instructed to drink in empty stomach, and to drink immediately after generation of water. The total amount that the patient drank the day before will be monitored by a researcher using survey form of mobile phone everyday.
  Other Names: Purified water (PW) generated from sham device

SUMMARY:
The goal of this clinical trial is to evaluate the effect of drinking electrolyzed alkaline reduced water (EARW) compared to drinking purified water (PW) on functional dyspepsia (FD) patients.

The main question[s] it aims to answer are:

* Drinking EARW (EARW group) will alleviate gastrointestinal (GI) symptoms and FD symptoms compared to drinking PW (PW group).
* Drinking EARW will make higher the FD-related Quality of Life (FD-QOL) compared to drinking PW.

Patients will drink EARW 10mL/kg/day body weight for 6 weeks according to the instruction of researcher using the experimental device installed at each patient's house. After 6 week, EARW and PW groups will be compared to evaluate effect of GI symptom and FD-related QOL.

DETAILED DESCRIPTION:
This study was designed as a randomized, parallel, double-blind controlled clinical trial. Enrolled patients with FD will be allocated randomly into two groups: EARW group and PW group. For 6 weeks, the patients will drink EARW and PW (10mL/kg/day body weight) in empty stomach condition. For the primary outcome measure, the gastrointestinal symptom rating scale (GSRS) will be used, and for the secondary outcome measure functional dyspepsia-related quality of life (FD-QoL), and Korean version of the Nepean Dyspepsia Index (NDI-K) will be used at baseline and at 6 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Symptoms onset should start at least 6 months before diagnosis based on one or more of the following symptoms Rome IV criteria (Unpleasant postprandial fullness, early satiety, epigastric pain, epigastric burning sensation)
* No evidence of structural disease in gastroscopy within the last 3 months
* Aged 19-70 years
* Who meets Rome IV criteria for functional dyspepsia
* Who have 4 or more symptoms based on the gastrointestinal symptom rating scale
* Patients who voluntarily agree to participate in this study and sign a written consent

Exclusion Criteria:

* Subjects who have a history of serious malignancy including gastrointestinal malignancy, cerebrovascular disease, and heart disease within the past 6 months were excluded

  * Subjects who have uncontrolled diabetes and hypertension despite appropriate management
  * Subjects who have a history of peptic ulcer or reflux esophagitis within the past 6 months were excluded
  * Subject who have history of gastrointestinal surgery were excluded
  * Women who are pregnant or breastfeeding
  * Subjects who are taking drugs that may affect the gastrointestinal tract (minimum of 2 weeks washout period is necessary before participating in the trial (Medications include H2 receptor blockers, anticholinergics, prostaglandins, proton pump inhibitors, gastromucosal protection agents, corticosteroids, non-steroidal anti-inflammatory drugs, aspirin, mucosal protective agents, etc.)
  * Subjects who are under drugs for therapeutic purposes such as functional food that promotes gastric health
  * Subjects who consumed more than 14 times alcohol per week in case of man and 7 times per week in case of female in the past 1 month

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2022-08-10 (Actual); Primary Completion 2022-10-28 (Actual); Study Completion 2022-11-29 (Actual)

PRIMARY OUTCOMES:
gastrointestinal symptom rating scale (GSRS) | 6 weeks
  The GSRS is a survey questionnaire designed to assess the symptoms associated with common GI disorders. It includes 15 questions on a scale of 1-7 that assess the inconvenience of the symptoms over the preceding period. A higher GSRS score indicates more inconvenient symptoms.

SECONDARY OUTCOMES:
functional dyspepsia-related quality of life (FD-QoL), | 6 weeks
  The FD-QoL questionnaire was used to measure the quality of life of FD patients. It includes total 21 items, and is categorized into 4: eating/diet (five items), daily activity (four items), emotion (six items), and social functioning (six items) on a 5-point Likert scale. A higher score indicates worse QoL.
Korean version of the Nepean Dyspepsia Index (NDI-K) | 6 weeks
  The NDI-K is a validated tool used for evaluating clinically meaningful FD changes, symptoms related to gastrointestinal problems. and it includes 15 symptom-based questions.
Inflammatory cytokines | 6 weeks
  Interleukin (IL)-1β, IL-10, IL-6, tumor necrosis factor (TNF)-α, and interferon gamma (IFN-γ) levels were measured to observe inflammatory immune response

CONTACTS AND LOCATIONS:
Overall Officials: Kyu-Jae Lee, Ph.D., Study Chair — 20, Ilsan-dong, Wonju, Gangwon-do, South Korea, 26426
Locations (1):
- Wonju Severance Christian Hospital, Wŏnju, Gwando, South Korea

IPD SHARING:
Plan to Share IPD: No